CLINICAL TRIAL: NCT05044624
Title: Retroperıtoneal Soft-Tıssue Sarcomas: Retrospectıve Clınıcal Study
Brief Title: Retroperıtoneal Soft-Tıssue Sarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mehmet acar, Investigator, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMU2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Retroperitoneal Sarcoma; Margin, Tumor-Free
Keywords: Soft tissue sarcoma; Surgery; Multidisciplinary Sarcoma Team
MeSH Terms: conditions — Margins of Excision; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Margin, Tumor-Free (Other)
  Interventions: Procedure: retroperitoneal mass excision

INTERVENTIONS:
Procedure: retroperitoneal mass excision — retroperitoneal mass excision

SUMMARY:
: Soft Tissue Sarcomas are rare mesenchymal tumors with many subtypes. Clean margin-wide resection is recommended for treatment. The guidelines recommend that sarcoma treatments be carried out in sarcoma centers. In this study, the location, histopathological features, clinical and demographic features, recurrence, and prognosis of retroperitoneal sarcomas were investigated.

DETAILED DESCRIPTION:
The demographic, histopathological, and immunohistochemical data of the patients who were operated on with the diagnosis of intraabdominal mass at Istanbul Medeniyet University Göztepe Prof. Dr. Süleyman Yalçın City Hospital from March 2016 to December 2020 were retrospectively evaluated. Ethical approval was obtained from Istanbul Medeniyet University Göztepe Prof. Dr. Süleyman Yalçın City Hospital Ethics Committee.

Patients diagnosed with pathological sarcoma subclass were included in the study. Patients younger than 18 years were excluded from the study. Visceral organ-origin sarcomas and extremity sarcomas were also excluded from the study. GIST's were included in sarcoma subtypes by WHO in 2013. However, they were not included in the study due to their solid organ origin.

The data of 18 patients' whore remained after the exclusion criteria were analyzed retrospectively. Pathology samples of the patients were re-examined by a single pathologist.

The demographic analysis was used for statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated with the diagnosis of intra-abdominal mass
* patients diagnosed with pathological sarcoma subclasses

Exclusion Criteria:

* Patients younger than 18 years
* Visceral organ-origin sarcomas
* extremity sarcomas
* GIST

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Clean margin wide resection | 63 month
  effect of clean surgical margin on recurrence

IPD SHARING:
Plan to Share IPD: Yes